CLINICAL TRIAL: NCT00496899
Title: Clinical Evaluation of New Computerized Labor Monitoring System.
Acronym: CLM
Status: Terminated | Type: Observational
Why Stopped: The study was stopped prematurally due to low recruiting
Sponsor: Barnev Ltd (Other)
Responsible Party: Clinical Trial Manager, Barnev
Other Study IDs: TASMC-07-AM-355-CITL
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2007-07

CONDITIONS: Obstetrics; Labor
Keywords: Labor; Obstetric; cervical dilatation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Women in active labor

SUMMARY:
The study is an open label feasibility study. The purpose of the study is to evaluate the ease of use of the Cervical ITR in terms of duration of attachment and number of detachments.

DETAILED DESCRIPTION:
Every year, millions of babies are born worldwide. Yet, despite great advances in medical technology, the method used to obtain the most critical parameter in labor management - cervix dilatation, remains a vaginal (manual) examination. This vaginal examination, intended to estimate the dilatation of the cervix and the progress of the baby's head, is inaccurate, non-continuous and involves the risk of infection to both fetus and mother. It is also uncomfortable to the mother. The consequences of infections or delayed treatment may range from simple complications to irreversible damage. Early detection of abnormal patterns of labor progress could prevent complications and shorten the labor process and hospitalization, thereby saving both aggravation and cost.

To truly manage the labor process, a labor management system is required. Such a system is expected to provide the obstetrical staff with the flow of accurate, continuous, real-time information, such as cervix dilatation.

ELIGIBILITY:
Inclusion Criteria:

* Laboring women referred to the Maternity Center in active labor (3cm dilatation and contractions).
* Gestational age 37-42 weeks. (GA)
* Single fetus
* Subjects who understood, agreed and signed the informed consent form

Exclusion Criteria:

* Women with abnormal placentation (placenta previa)
* Women with coagulation abnormalities.
* Abnormal fetal presentation (breech presentation)
* Maternal History of HIV and/or blood transmitted hepatitis and/or active genital Herpes.
* Preterm premature rupture of membranes.
* Need for immediate delivery (cord prolapsed or suspected placental abruption

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Laboring women reffered to maternity center in active labor (3 -7 cm)dilatation and contraction
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Many, MD, Principal Investigator — Sackler school of medicine, Tel Aviv University
Locations (1):
- Tel Aviv soraski medical center, Tel Aviv, Israel